CLINICAL TRIAL: NCT01910818
Title: Understanding and Reversing Chronic Radiation Dermatitis - A Pilot Study
Brief Title: Pilot Study of the Effect of Laser on Reversing Chronic Radiation Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Director, Wellman Center for Photomedicine, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2013P000988
Record Dates: First submitted 2013-06-05; First posted 2013-07-30 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Chronic Radiation Dermatitis
Keywords: radiation; dermatitis; laser; fractional; CO2; chronic; fibrosis; scar
MeSH Terms: conditions — Dermatitis; Bronchiolitis Obliterans Syndrome; Fibrosis; Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fractional CO2 laser Treatment (Experimental): This is the area getting treated with CO2 laser.
  Interventions: Device: Fractional CO2 laser treatment
- No Treatment (Experimental): This is the area receiving no treatment.
  Interventions: Other: No treatment

INTERVENTIONS:
Device: Fractional CO2 laser treatment — Patient will be treated with fractional laser treatment over the areas with fibrosis.
  Other Names: Lumenis Ultrapulse CO2 laser
  Arms: Fractional CO2 laser Treatment
Other: No treatment — Patient will also have an area that is not being treated with CO2 laser. This is the area not getting treatment.
  Arms: No Treatment

SUMMARY:
Radiotherapy, an essential modality in cancer treatment, frequently induces a fibrotic process in the skin which can lead to increased risk of malignancy, poor wound healing, pain and limitation of movement, and permanent loss of skin appendages with hyper/hypopigmentation, decreased sweating and xerosis, posing significant cosmetic and quality of life issues. Advances in laser therapy has led to the use of fractional laser treatment (FLT) to treat fibrosis associated with in hypertrophic scars and morphea, leading to tissue repair, scar remodeling. The investigators propose a pilot clinical study to test the hypothesis that FLT can normalize the fibrotic process and induce normal scar remodeling in patients affected by chronic radiation injury. Understanding and correcting this underlying fibrotic process can help restore normal skin functions in patients affected with chronic radiation dermatitis (RD) and other debilitating fibrotic diseases in dermatology such as scleroderma, morphea, or nephrogenic systemic fibrosis.

DETAILED DESCRIPTION:
We propose to treat 22 patients with significant radiation induced fibrosis (RIF) and skin changes. Each patient will receive fractional treatment (FLT) using the Lumenis Ultrapulse Carbon Dioxide (CO2) laser as well as control (no treatment) randomized to site. Patient age, type of cancer, method/dosage of radiation, latency between radiation treatment and start of study, and characteristics of skin changes will be recorded, including fibrosis surface area, depth, color, and compliance. Assessments will be conducted before each treatment, after each treatment, and 3-12 months after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females between 18 and 80 years of age with radiation-induced fibrosis and depigmentation. The fibrosis must have occurred at least 1 year prior to the date of enrollment.
2. Having suitable areas of treatment: All wounds in the area of interest must be closed for at least two months. The scars must be deemed stable for a period of 3 months or have a suitable contralateral control before initiation of treatment. This will be determined by objective measurements of scar erythema, pliability, induration, thickness at enrollment and again at 3 months;
3. Fitzpatrick skin types I-VI;
4. Able and willing to comply with all visit, treatment and evaluation schedules and requirements;
5. Able to understand and provide written informed consent;
6. Pregnant woman can be included because study involves local intervention, no new drugs.

Exclusion Criteria:

1. Active tanning, including the use of tanning booths, during the course of the study;
2. Prior skin treatment with laser or other devices in the treated area within three months of initial treatment or during the course of the study;
3. Adverse reactions to compounds of any external agent (e.g., gels, lotions or anesthetic creams) required for use in the study, if no alternative to the said agent exists;
4. History of collagen vascular disease;
5. Active Herpes Simplex or Zoster at the time of treatment or having experienced more than three episodes of Herpes Simplex / Zoster eruption within a year of study enrollment;
6. History of immunosuppression/immune deficiency disorders (including human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS) or use of immunosuppressive medications;
7. Having any form of active cancer at the time of enrollment and during the course of the study;
8. Significant concurrent illness, such as uncontrolled diabetes (with a hemoglobin A1C of more than 8) (i.e., any disease state that in the opinion of the Investigator would interfere with the anesthesia, treatment, or healing process); Mentally incompetent, prisoner or evidence of active substance or alcohol abuse;
9. Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or study personnel) to treat the subject as part of this research study;
10. If it is determined that the contracture is due to a deeper process involving the muscles, ligaments or bones.
11. Patient on chemotherapy (but not tamoxifen or other things that affect wound healing) and also active XRT
12. Participation in another interventional study with potential exposure to an investigational drug within past 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-11; Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Improvement in fibrosis (% reduction in fibrosis surface area) compared to controlled sites | 6-12 months
  The primary end point is % reduction of the fibrosis surface area compared to control sites at 6-12 months.

SECONDARY OUTCOMES:
Adverse events | 2 years
  Measurement adverse events (infection, scarring, ulceration, excessive bleeding, poor wound healing)

CONTACTS AND LOCATIONS:
Overall Officials: Richard R Anderson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Wellman Center for Photomedicine, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: clinical trials — https://rally.partners.org/study/chronic_radiation_dermatitis